CLINICAL TRIAL: NCT00395629
Title: A Phase I/II Open Label, Dose Escalation Trial and a Six Month Extension to Explore the Safety and Efficacy of ICL670 in Patients With Iron Overload Resulting From Hereditary Hemochromatosis.
Brief Title: Safety and Efficacy of Deferasirox (ICL670) in Patients With Iron Overload Resulting From Hereditary Hemochromatosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670A2202; EudraCT no. 2006-002102-57 (Registry Identifier: EudraCT)
Record Dates: First submitted 2006-11-01; First posted 2006-11-03 (Estimated); Results first posted 2011-05-18 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Iron Overload; Hereditary Hemochromatosis
Keywords: Deferasirox; ICL670A; Iron chelators; Deferiprone; Transfusional Hemochromatosis
MeSH Terms: conditions — Iron Overload; Hemochromatosis | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ICL670 (Deferasirox) (Experimental): Three dose cohorts: 5 mg/kg/day, 10 mg/kg/day, 15 mg/kg/day
  Interventions: Drug: Deferasirox (ICL670)

INTERVENTIONS:
Drug: Deferasirox (ICL670)

SUMMARY:
Brief Summary: This study was designed to explore a safe dose and characterize the preliminary safety and efficacy of ICL670 in adult patients with previously documented history of homozygous C282Y.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age or older
* Male or female patients homozygous for the C282Y mutation.
* Iron overload as documented by serum ferritin and transferrin saturation
* No known allergy or contraindication to the administration of deferasirox
* Ability to comply with all study-related procedures, medications, and evaluations
* Effective use of birth control measures.

Exclusion Criteria:

* Iron overload not due to hereditary hemochromatosis
* Males with hemoglobin <13 mg/dL, females with hemoglobin <12 mg/dL
* Desferal treatment within 1 month of the screening visit
* Patients currently or previously treated with deferiprone or deferasirox
* Significant medical condition interfering with the ability to partake in this study
* Presence of a surgical or medical condition that might significantly alter the absorption, distribution, metabolism or excretion of any study drug
* Clinical evidence of Active Hepatitis B or C
* Positive HIV serology
* Pregnant or breast feeding patients
* Patients treated with systemic investigational drug within 4 weeks prior or with topical investigational drug within 7 days prior to the screening visit

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2006-08; Primary Completion 2007-12 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, M.D., Study Director — Novartis Pharmaceuticals
Locations (18):
- United States (9):
  - UC Irvine/Long Beach, Long Beach, California
  - University of Connecticut Health Center, Farmington, Connecticut
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - St. Louis University, St Louis, Missouri
  - Rochester General Hospital, Rochester, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Three Medical Park, Columbia, South Carolina
- Novartis Investigative Site, Brisbane, Australia
- Novartis Investigative Site, London, Ontario, Canada
- Novartis Investigative Site, Rennes, France
- Germany (4):
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Oberhausen
- Italy (2):
  - Novartis Investigative Site, Modena
  - Novartis Investigative Site, Monza

REFERENCES:
- See also: Related Info — http://www.novartisclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Deferasirox (ICL670) 5 mg/kg/Day; Deferasirox (ICL670) 10 mg/kg/Day; Deferasirox (ICL670) 15 mg/kg/Day: Deferasirox (ICL670) was provided as 125 mg, 250 mg, and 500 mg tablets. Dosage was based on the participant's body weight. ICL670 was administered orally, once a day, 30 minutes prior to breakfast.
Period: Core Study
Arm/Group | Deferasirox (ICL670) 5 mg/kg/Day | Deferasirox (ICL670) 10 mg/kg/Day | Deferasirox (ICL670) 15 mg/kg/Day
Started | 11 | 15 | 23
Completed | 10 | 11 | 16
Not Completed | 1 | 4 | 7
Not completed — Adverse Event | 0 | 3 | 4
Not completed — Abnormal laboratory value(s) | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Period: Extension Study
Arm/Group | Deferasirox (ICL670) 5 mg/kg/Day | Deferasirox (ICL670) 10 mg/kg/Day | Deferasirox (ICL670) 15 mg/kg/Day
Started | 9 | 6 | 11
Completed | 9 | 6 | 8
Not Completed | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Administrative problems | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deferasirox (ICL670) 5 mg/kg/Day | Deferasirox (ICL670) 10 mg/kg/Day | Deferasirox (ICL670) 15 mg/kg/Day | Total
Number analyzed (Participants) | 11 | 15 | 23 | 49
Age Continuous [Mean (Standard Deviation); unit: years] — The n values in the Extension Study Category are the number of participants in each Arm/Group. The last n value= 26 is the Total number of participants.
  years
    Core Study | 55.8 (12.78) | 47.8 (10.26) | 49.8 (16.41) | 50.6 (14.04)
    Extension Study (n=9,6,11,26) | 55.7 (14.23) | 44.8 (10.61) | 50.1 (15.88) | 50.8 (14.34)
Sex/Gender, Customized [Number; unit: participants]
  Female_Core Study | 2 | 4 | 10 | 16
  Male_Core Study | 9 | 11 | 13 | 33
Sex/Gender, Customized [Number; unit: participants]
  Female_Extension Study | 1 | 1 | 3 | 5
  Male_Extension Study | 8 | 5 | 8 | 21
  Core Participants not enrolled in the Extension | 2 | 9 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change of Serum Ferritin From Baseline to the End of Extension, by Dose Cohort (Extension Per-protocol Population)
Description: Mean absolute change in serum ferritin from baseline to the end of the extension study.
Time Frame: 0 to 48 weeks
Population: Extension Per-protocol population including all participants of the per protocol population who also were part of the extension safety population.
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Deferasirox (ICL670) 5 mg/kg/Day | Deferasirox (ICL670) 10 mg/kg/Day | Deferasirox (ICL670) 15 mg/kg/Day
Number analyzed (Participants) | 9 | 6 | 11
µg/L | -389.1 (185.35) | -610.5 (341.84) | -571.6 (552.81)

2. Secondary Outcome: Trough Concentrations of Deferasirox (ICL670), by Dose Cohort (Per-protocol Population)
Description: A blood sample was collected just prior to administration of the next dose of Deferasirox (pre-dose trough level) or approximately 24 hours after the previous dose at weeks 4, 8, 12, 16, 20 and 24. The mean trough concentration at each time point was calculated.
Time Frame: 4, 8, 12, 16, 20, and 24 weeks
Population: Per-protocol population included all participants of the safety population; who received at least one dose of study drug within the core study and had at least one safety assessment, and who did not have any major protocol deviation. n in each of the Categories is the number of participants in each arm/group who had data for that time point.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Deferasirox (ICL670) 5 mg/kg/Day | Deferasirox (ICL670) 10 mg/kg/Day | Deferasirox (ICL670) 15 mg/kg/Day
Number analyzed (Participants) | 11 | 15 | 22
µmol/L
  Week 4 (n=10,14,17) | 9.63 (8.783) | 19.62 (9.502) | 30.48 (20.201)
  Week 8 (n=10,12,17) | 8.86 (5.828) | 23.88 (22.787) | 27.06 (21.686)
  Week 12 (n=10,12,13) | 10.58 (11.752) | 28.71 (23.849) | 23.39 (11.403)
  Week 16 (n=10,11,11) | 12.38 (11.634) | 21.62 (16.539) | 21.80 (18.713)
  Week 20 (n=9,10,8) | 11.72 (10.316) | 26.47 (17.934) | 27.58 (25.324)
  Week 24 (n=10,9,6) | 14.62 (12.216) | 21.32 (21.840) | 26.83 (11.178)

ADVERSE EVENTS:
Description: Safety Population includes all participants who received at least one dose of study drug and had at least one safety assessment.
Groups:
- Deferasirox (ICL670) 5 mg/kg/day_Core Study; Deferasirox (ICL670) 10 mg/kg/day_Core Study; Deferasirox (ICL670) 15 mg/kg/day_Core Study; Deferasirox (ICL670) 5 mg/kg/day_Extension Study; Deferasirox (ICL670) 10 mg/kg/day_Extension Study; Deferasirox (ICL670) 15 mg/kg/day_Extension Study: Deferasirox (ICL670) was provided as 125 mg, 250 mg, and 500 mg tablets. Dosage was based on the participant's body weight. ICL670 was administered orally, once a day, 30 minutes prior to breakfast.
Arm/Group | Deferasirox (ICL670) 5 mg/kg/day_Core Study | Deferasirox (ICL670) 10 mg/kg/day_Core Study | Deferasirox (ICL670) 15 mg/kg/day_Core Study | Deferasirox (ICL670) 5 mg/kg/day_Extension Study | Deferasirox (ICL670) 10 mg/kg/day_Extension Study | Deferasirox (ICL670) 15 mg/kg/day_Extension Study
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/15 | 0/23 | 1/9 | 0/6 | 0/11
Other Adverse Events (participants affected / at risk) | 10/11 | 14/15 | 23/23 | 9/9 | 5/6 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Deferasirox (ICL670) 5 mg/kg/day_Core Study (N=11) | Deferasirox (ICL670) 10 mg/kg/day_Core Study (N=15) | Deferasirox (ICL670) 15 mg/kg/day_Core Study (N=23) | Deferasirox (ICL670) 5 mg/kg/day_Extension Study (N=9) | Deferasirox (ICL670) 10 mg/kg/day_Extension Study (N=6) | Deferasirox (ICL670) 15 mg/kg/day_Extension Study (N=11)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Deferasirox (ICL670) 5 mg/kg/day_Core Study (N=11) | Deferasirox (ICL670) 10 mg/kg/day_Core Study (N=15) | Deferasirox (ICL670) 15 mg/kg/day_Core Study (N=23) | Deferasirox (ICL670) 5 mg/kg/day_Extension Study (N=9) | Deferasirox (ICL670) 10 mg/kg/day_Extension Study (N=6) | Deferasirox (ICL670) 15 mg/kg/day_Extension Study (N=11)
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 2 | 1 | 0 | 0
Mixed deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neurosensory hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 2 | 0 | 0
Blindness day (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 1
Corneal opacity (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Maculopathy (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Presbyopia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 4 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 6 | 10 | 2 | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 2 | 1
Flatulence (Gastrointestinal disorders) | 2 | 1 | 2 | 1 | 0 | 2
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1 | 0
Gingival disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 6 | 0 | 0 | 4
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 2
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 2 | 2 | 1 | 1
Influenza like illness (General disorders) | 0 | 1 | 2 | 0 | 1 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 0 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1 | 3 | 1 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 3
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 3 | 3 | 1 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 3 | 4 | 1 | 2 | 3
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Creatinine renal clearance decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Creatinine renal clearance increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 1 | 2 | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 1 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 2 | 3 | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 2 | 7 | 1 | 0 | 5
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Syncope vasovagal (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 2 | 1 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 3
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 4 | 1 | 1 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.